CLINICAL TRIAL: NCT05318261
Title: Incidence of Weaning-induced Pulmonary Oedema (The WIPO Study)
Brief Title: Incidence and Risk Factors of Weaning-induced Cardiac Dysfunction: Results From a Multicenter, Observational Study
Acronym: WIPO
Status: Completed | Type: Observational
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Principal Investigator, Bicetre Hospital
Other Study IDs: 2017-A00392-51
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Weaning Failure; Weaning-induced Pulmonary Edema; Spontaneous Breathing Trial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Spontaneous breathing trial — A spontaneous breathing trial (SBT) is used to identify patients who are likely to fail liberation from mechanical ventilation. The test can be done according to the usual modalities of the participating centre, following the international recommendations, meaning either by disconnecting the endotracheal tube from the ventilator and connecting it to a source of oxygen through the T-tube or by setting pressure support with low positive end-expiratory pressure (PEEP). The choice of the method will not be determined according to the participation in this study but will be done according to the habits of the participating centre.

SUMMARY:
During weaning from mechanical ventilation, the shift from positive to negative pressure ventilation may be responsible for a cardiac dysfunction that can lead to the development of pulmonary oedema (weaning-induced pulmonary oedema, WIPO) and to the failure of spontaneous breathing trials. However, the incidence and risk factors for WIPO development are not well defined and have been investigated only by a few studies.

DETAILED DESCRIPTION:
During weaning from mechanical ventilation, the shift from positive to negative pressure ventilation may be responsible for a cardiac dysfunction that can lead to the development of pulmonary oedema (weaning-induced pulmonary oedema, WIPO) and to the failure of spontaneous breathing trials. The mechanisms leading to WIPO have been described in many studies. The fact that the intrathoracic pressure becomes negative increases right ventricle preload and afterload, reduces right ventricle compliance and increases left ventricle afterload. Arterial hypertension, which results from adrenergic stress and possibly from hypercapnia, usually worsens this latter mechanism. Myocardial ischemia, resulting from the imbalance between the reduction of oxygen delivery (hypoxemia) and increased oxygen demand (unfavourable loading conditions, increase of inotropic and heart rate) may participate in this phenomenon, even though its incidence seems to be low. The means for detecting WIPO in a patient performing a spontaneous breathing trial (SBT) have been widely investigated. To avoid the insertion of a pulmonary artery catheter, which clinicians nowadays tend to avoid when the patient is ready to be extubated, many alternatives methods have been proposed. The increase of left ventricular filling pressure during an SBT was detected with echocardiography, the increase during the test either of B-type natriuretic peptide levels or of extravascular lung water measured by transpulmonary thermodilution can be used. The investigators have also demonstrated that the detection of haemoconcentration during a weaning test, which is related to the filtration of a significant amount of plasma through the alveolar-capillary barrier, allows the detection of WIPO.

Unresolved questions:

The incidence of WIPO is not well defined. In the studies where it has been reported, it ranged between 44% and 87% of SBT failures. However, these studies included a small number of patients and/or included a specific population of patients that had already failed one or more weaning tests. In a monocentric study, the investigators recently reported that WIPO occurred in 59% of cases of SBT failures.

The risk factors for WIPO development are not well defined and have been investigated only by a few studies. In the above-mentioned one, the investigators have identified the presence of pre-existing cardiopathy, pre-existing chronic respiratory failure and obesity as independent risk factors for developing WIPO. However, these results were obtained only from a monocentric cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Social coverage from health insurance (in France).
3. Decision of the attending physicians to perform an SBT.

Exclusion Criteria:

1. Presence of tracheostomy (in this case at the end of the test the patient could be connected to the ventilator, even in case of positivity of the weaning test. Thus, it is not possible to test the absence of reintubation at 48 hours, which is one of the criteria defining the success of weaning).
2. Refusal of the patient or, if the case, one of the relatives to participate to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the intubated patients who need to do a Spontaneous Breathing Trial
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
The incidence of WIPO | 30-120 mins during the Spontaneous Breathing Trial
  The diagnosis of WIPO will be done a posteriori by a group of experts. They will establish the diagnosis of WIPO, based on the following elements:
  * Failure or success of SBT
  * Clinical examination at the end of SBT
  * Variation during SBT of arterial blood gas variables, plasmatic protein and blood haemoglobin concentration, extravascular lung water (optional), B-type natriuretic peptide (optional), echocardiographic estimation of left ventricular preload (E and A waves of mitral flow, e' wave of the mitral valve annulus), pulmonary arterial occlusion pressure (optional).

SECONDARY OUTCOMES:
Risk factors for developing WIPO | The risk factors for WIPO will be done a posteriori by multivaraite analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dres M, Teboul JL, Monnet X. Weaning the cardiac patient from mechanical ventilation. Curr Opin Crit Care. 2014 Oct;20(5):493-8. doi: 10.1097/MCC.0000000000000131. PMID 25159477
- [Result] Teboul JL. Weaning-induced cardiac dysfunction: where are we today? Intensive Care Med. 2014 Aug;40(8):1069-79. doi: 10.1007/s00134-014-3334-4. Epub 2014 May 27. PMID 24861350
- [Result] Lemaire F, Teboul JL, Cinotti L, Giotto G, Abrouk F, Steg G, Macquin-Mavier I, Zapol WM. Acute left ventricular dysfunction during unsuccessful weaning from mechanical ventilation. Anesthesiology. 1988 Aug;69(2):171-9. doi: 10.1097/00000542-198808000-00004. PMID 3044189
- [Result] Liu J, Shen F, Teboul JL, Anguel N, Beurton A, Bezaz N, Richard C, Monnet X. Cardiac dysfunction induced by weaning from mechanical ventilation: incidence, risk factors, and effects of fluid removal. Crit Care. 2016 Nov 12;20(1):369. doi: 10.1186/s13054-016-1533-9. PMID 27836002
- [Result] Lamia B, Maizel J, Ochagavia A, Chemla D, Osman D, Richard C, Teboul JL. Echocardiographic diagnosis of pulmonary artery occlusion pressure elevation during weaning from mechanical ventilation. Crit Care Med. 2009 May;37(5):1696-701. doi: 10.1097/CCM.0b013e31819f13d0. PMID 19325473
- [Result] Grasso S, Leone A, De Michele M, Anaclerio R, Cafarelli A, Ancona G, Stripoli T, Bruno F, Pugliese P, Dambrosio M, Dalfino L, Di Serio F, Fiore T. Use of N-terminal pro-brain natriuretic peptide to detect acute cardiac dysfunction during weaning failure in difficult-to-wean patients with chronic obstructive pulmonary disease. Crit Care Med. 2007 Jan;35(1):96-105. doi: 10.1097/01.CCM.0000250391.89780.64. PMID 17095948
- [Result] Dres M, Teboul JL, Anguel N, Guerin L, Richard C, Monnet X. Extravascular lung water, B-type natriuretic peptide, and blood volume contraction enable diagnosis of weaning-induced pulmonary edema. Crit Care Med. 2014 Aug;42(8):1882-9. doi: 10.1097/CCM.0000000000000295. PMID 24717458
- [Result] Perren A, Domenighetti G, Mauri S, Genini F, Vizzardi N. Protocol-directed weaning from mechanical ventilation: clinical outcome in patients randomized for a 30-min or 120-min trial with pressure support ventilation. Intensive Care Med. 2002 Aug;28(8):1058-63. doi: 10.1007/s00134-002-1353-z. Epub 2002 Jul 13. PMID 12185425
- [Result] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Result] Cabello B, Thille AW, Roche-Campo F, Brochard L, Gomez FJ, Mancebo J. Physiological comparison of three spontaneous breathing trials in difficult-to-wean patients. Intensive Care Med. 2010 Jul;36(7):1171-9. doi: 10.1007/s00134-010-1870-0. Epub 2010 Mar 30. PMID 20352189
- [Result] Dres M, Teboul JL, Anguel N, Guerin L, Richard C, Monnet X. Passive leg raising performed before a spontaneous breathing trial predicts weaning-induced cardiac dysfunction. Intensive Care Med. 2015 Mar;41(3):487-94. doi: 10.1007/s00134-015-3653-0. Epub 2015 Jan 24. PMID 25617264
- [Result] Caille V, Amiel JB, Charron C, Belliard G, Vieillard-Baron A, Vignon P. Echocardiography: a help in the weaning process. Crit Care. 2010;14(3):R120. doi: 10.1186/cc9076. Epub 2010 Jun 22. PMID 20569504
- [Derived] Shi R, Ayed S, Beuzelin M, Persichini R, Legouge M, Vita NDE, Levy B, Beurton A, Mangal K, Hullin T, Labbe V, Guillot M, Harrois A, Cecconi M, Anguel N, Osman D, Moretto F, Lai C, Pham T, Teboul JL, Monnet X. Incidence and risk factors of weaning-induced pulmonary oedema: results from a multicentre, observational study. Crit Care. 2025 Mar 31;29(1):140. doi: 10.1186/s13054-025-05350-6. PMID 40165223